CLINICAL TRIAL: NCT04902911
Title: Point of Care Evaluation of Novir 2019-nCoV Immunoglobulin G/ Immunoglobulin M (IgG/IgM) Antibody Test (Collodial Gold)
Acronym: NOVIR POC
Status: Terminated | Type: Observational
Why Stopped: Failed to meet FDA criteria on one target at FDA, CDC, and market is not looking for rapid antibody tests.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Novir (Unknown)
Responsible Party: Principal Investigator, Matthew Faron, PhD, Assistant Professor of Pathology, Medical College of Wisconsin
Other Study IDs: PRO00039709
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Covid19
Keywords: covid 19; antibody; IgM; IgG
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Antigen testing in those who have history of COVID-19: Individuals must have had history of COVID-19. Finger stick point of care test will be performed which results in 10 minutes indicating if there is detection of a control, IgG and IgM. Control line must be present for test to be considered valid. 3mL of venous whole blood will be collected from patient in which the research team will perform the SARS-CoV-2 antibody test.
  Interventions: Device: COVID-19 SARS-CoV IgG/IgM antibody rapid test
- Antigen testing in those who do not have history of COVID-19 and COVID immunization: Individuals may not have history of COVID-19 and COVID immunizations in order to be eligible. Finger stick point of care test will be performed which results in 10 minutes indicating if there is detection of a control, IgG and IgM. Control line must be present for test to be considered valid. 3mL of venous whole blood will be collected from patient in which the research team will perform the SARS-CoV-2 antibody test.
  Interventions: Device: COVID-19 SARS-CoV IgG/IgM antibody rapid test

INTERVENTIONS:
Device: COVID-19 SARS-CoV IgG/IgM antibody rapid test — Needle stick point of care and 3mL vial of blood will be collected and tested for individual without history of COVID-19 and immunization as well as a second group composed of individuals with history of COVID-19

SUMMARY:
This clinical study is designed to test the efficacy of the Novir 2019-nCoV Immunoglobulin M/Immunoglobulin G Antibody Test in a point-of-care setting to support the increasing need for rapid screening in the detection of antibodies. The study is performed on individuals who have no history of COVID-19 and no history of COVID immunization as well as individuals with history of COVID-19 that was diagnosed greater than 15 days. This is performed both through 3mL venous whole blood which is ran through an assay as well a point-of-care rapid test which is resulted in 10 minutes. Aiding in the rapid detection of COVID-19 antibodies.

DETAILED DESCRIPTION:
This clinical study is designed to test the efficacy and robustness of the Novir 2019-nCoV IgM/IgG Antibody Test (Colloidal Gold) in a point-of-care (POC) setting to support the growing need for rapid screening of patients to detect antibodies. The COVID-19 SARS-CoV IgM/IgG antibody rapid test is an immunochromatographic lateral flow assay intended for qualitative detection of IgM and IgG antibodies to SARS-CoV-2 in human venipuncture and finger stick whole blood. The COVID-19 SARS-CoV IgM/IgG antibody rapid test is intended for use as an aid in identifying individuals with an adaptive immune response to SARS-CoV-2, indicating recent or prior infection. At this time, it is unknown for how long antibodies persist following infection and if the presence of antibodies confers protective immunity.

Results are for the detection of SARS CoV-2 antibodies. IgM and IgG antibodies to SARS-CoV-2 are generally detectable in blood several days after initial infection, although the duration of time antibodies are present post-infection is not well characterized. Individuals may have detectable virus present for several weeks following seroconversion. All the results will be compared to an FDA EUA authorized PCR test results and may also be compared to an FDA EUA authorized ELISA, CMIA, or other antibody test.

The study results will be used for an EUA application to the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Must be 21 years old or older.
* Must be able to provide finger stick and venous whole blood samples.
* Must be able to understand and sign a consent form.
* Must be able to provide an additional sample(s) required by the study site for an additional FDA EUA authorized antibody testing (ELISA, CMIA, or other antibody test).
* Has an immediate need to determine COVID-19 status for occupational purposes.
* Was exposed to a COVID-19 patient within 7 days that leads the healthcare provider to suspect the individual of possibly having SARS-CoV-2 infection.
* Has symptoms that lead the healthcare provider to suspect the individual of possibly having SARS-CoV-2 infection.
* Has had a positive FDA EUA authorized PCR test between 1-28 days with or without symptom expression.
* Individuals who have tested positive for COVID-19 infection and have antibodies detected must have agreed to participate in the MCW Tissue Bank COVID-19 banking project.

Exclusion Criteria:

* Is receiving treatment with infusion of convalescent plasma or other antibody therapy related to SARS-CoV-2 infections.
* Tested negative for COVID-19 by PCR more than 7 days ago.
* Is participating in a SARS-CoV-2 vaccine study.or received any doses of the available SARS-CoV-2 vaccines.
* Previously tested positive for COVID-19 at any point in time (for asymptomatic patients enrolling in the negative patient population).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any subject willing to participate since status for previous infection is not needed.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Novir 2019-nCoV IgG/IgM Antibody test | 2 years
  To determine the sensitivity and specificity of the Novir 2019-nCoV IgM/IgG Antibody Test (Colloidal Gold) when testing intended use populations who meet the criteria of having COVID-19 infection by Centers for Disease Control and Prevention (CDC). The test is to be performed by healthcare professionals (non-CLIA laboratory technicians) at POC settings.vStandard calculations will be used to derive sensitivity, specificity, positive and negative predictive values as well as 95% confidence intervals compared to reference method.

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Health WAC, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No